CLINICAL TRIAL: NCT02366689
Title: Clinical Efficacy in Reducing Established Dental Plaque and Gingivitis of a Toothpaste Containing 0.3% Triclosan, 2% Copolymer / Sodium Fluoride and a Manual Toothbrush as Compared to an Oral Hygiene Multi-component Regimen Encompassing the Use of a Manual Toothbrush, a Toothpaste Containing Stannous Fluoride / Sodium Hexametaphosphate and a Mouthwash Containing 0.07% Cetylpyridinium Chloride
Brief Title: Clinical Study Comparing Dental Plaque and Gingivitis Reduction After Using One of Three Oral Hygiene Multi-component Regimens (Using of a Manual Toothbrush, a Toothpaste and a Mouthwash)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2014-05-PG-6MCTCPG-ED
Record Dates: First submitted 2015-02-06; First posted 2015-02-19 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2015-02

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Toothpaste (Active Comparator): Triclosan/fluoride toothpaste
  Interventions: Drug: Triclosan/fluoride toothpaste
- Toothpaste + mouthwash (Active Comparator): stannous fluoride toothpaste + cetylpyridinium chloride Mouthwash
  Interventions: Drug: stannous fluoride toothpaste; Drug: Cetylpyridinium chloride mouthwash
- Fluoride only Toothpaste + mouthwash (Placebo Comparator): Fluoride only toothpaste + Fluoride only Mouthwash
  Interventions: Drug: fluoride only toothpaste; Drug: Fluoride only mouthwash

INTERVENTIONS:
Drug: Triclosan/fluoride toothpaste — Brush whole mouth with Total toothpaste (triclosan/fluoride) using Total 360 toothbrush for 1 minute, 2 times/day for 6 months (study duration).
  Other Names: Total toothpaste
  Arms: Toothpaste
Drug: stannous fluoride toothpaste — Brush whole mouth with Crest Pro-Health toothpaste using an Oral B Pro-Health toothbrush for 1 minute, 2 times/day for 6 months (study duration).
  Other Names: Crest Pro-Health toothpaste
  Arms: Toothpaste + mouthwash
Drug: fluoride only toothpaste — Brush whole mouth with Crest Cavity Protection toothpaste using an Oral B Indicator toothbrush for 1 minute, 2 times/day for 6 months (study duration). Immediately after each brushing, rinse whole mouth with 20 ml of Crest fluoride Mouthwash for 30 seconds.
  Other Names: Crest Cavity Protection toothpaste
  Arms: Fluoride only Toothpaste + mouthwash
Drug: Cetylpyridinium chloride mouthwash — Immediately after each brushing with Crest Pro-Health toothpaste, rinse whole mouth with 20 ml of Crest Pro-Health Mouthwash for 30 seconds.
  Other Names: Crest Pro-Health Multi-Protection Mouthwash
  Arms: Toothpaste + mouthwash
Drug: Fluoride only mouthwash — Immediately after each brushing with Crest Cavity Protection toothpaste, rinse whole mouth with 20 ml of Crest Pro-Health For Me mouthwash for 30 seconds.
  Other Names: Crest Pro-Health For Me Breezy Mint mouthwash
  Arms: Fluoride only Toothpaste + mouthwash

SUMMARY:
The objective of this clinical research study is to assess the efficacy of a commercially available triclosan/copolymer toothpaste compared to a commercially available oral hygiene multi-component regimen encompassing the use of a manual toothbrush, a toothpaste containing stannous fluoride / sodium hexametaphosphate and a mouthwash containing cetylpyridinium chloride relative to a negative control regimen in reducing established dental plaque and gingivitis over three and six months of assigned product use.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ages 18-70, inclusive.
2. Availability for the six-month duration of the study.
3. Good general health.
4. Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
5. Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
6. Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
7. Signed Informed Consent Form.

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial removable dentures.
3. Tumor(s) of the soft or hard tissues of the oral cavity.
4. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
5. Five or more carious lesions requiring immediate restorative treatment.
6. Use of antibiotics any time during the one month prior to entry into the study.
7. Participation in any other clinical study or test panel within the one month prior to entry into the study.
8. Pregnant women or women who are breast feeding.
9. Dental prophylaxis received in the past two weeks prior to baseline examinations.
10. History of allergies to oral care/personal care consumer products or their ingredients.
11. On any prescription medicines that might interfere with the study outcome.
12. An existing medical condition which prohibits eating or drinking for periods up to 4 hours.
13. History of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia Clinical Research, Cedar Knolls, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment of subjects is done locally by the clinical site
Pre-assignment Details: No washout or pre-assignment phase
Period: Overall Study
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Started | 60 | 58 | 61
Completed | 56 | 55 | 59
Not Completed | 4 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Pregnancy | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash | Total
Number analyzed (Participants) | 60 | 58 | 61 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.09 (11.72) | 48.65 (12.84) | 48.51 (12.90) | 49.08 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 47 | 146
  Male | 13 | 6 | 14 | 33
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 61 | 179

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Scores
Description: Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Number analyzed (Participants) | 60 | 58 | 61
units on a scale | 3.33 (0.28) | 3.22 (0.27) | 3.34 (0.26)
Statistical Analysis 1: Comparison: Toothpaste vs Toothpaste + Mouthwash vs Fluoride Only Toothpaste + Mouthwash; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.04, ANOVA

2. Primary Outcome: Dental Plaque Scores
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Number analyzed (Participants) | 56 | 57 | 59
units on a scale | 2.26 (0.23) | 2.42 (0.22) | 2.66 (0.23)
Statistical Analysis 1: Comparison: Toothpaste vs Toothpaste + Mouthwash vs Fluoride Only Toothpaste + Mouthwash; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Primary Outcome: Dental Plaque Scores
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Number analyzed (Participants) | 56 | 55 | 59
units on a scale | 1.84 (0.25) | 1.86 (0.29) | 2.37 (0.32)
Statistical Analysis 1: Comparison: Toothpaste vs Toothpaste + Mouthwash vs Fluoride Only Toothpaste + Mouthwash; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Primary Outcome: Gingivitis Scores
Description: Gingivitis scale (Loe & Silness Gingival Index) Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Number analyzed (Participants) | 60 | 58 | 61
units on a scale | 2.18 (0.16) | 2.17 (0.22) | 2.22 (0.21)
Statistical Analysis 1: Comparison: Toothpaste vs Toothpaste + Mouthwash vs Fluoride Only Toothpaste + Mouthwash; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.432, ANOVA

5. Primary Outcome: Gingivitis Scores
Description: as for outcome 4
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Number analyzed (Participants) | 56 | 56 | 59
units on a scale | 1.48 (0.15) | 1.65 (0.16) | 1.89 (0.17)
Statistical Analysis 1: Comparison: Toothpaste vs Toothpaste + Mouthwash vs Fluoride Only Toothpaste + Mouthwash; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Primary Outcome: Gingivitis Scores
Description: as for outcome 4
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Number analyzed (Participants) | 56 | 55 | 59
units on a scale | 1.17 (0.14) | 1.18 (0.12) | 1.85 (0.13)
Statistical Analysis 1: Comparison: Toothpaste vs Toothpaste + Mouthwash vs Fluoride Only Toothpaste + Mouthwash; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline, 3 months and 6 months
Arm/Group | Toothpaste | Toothpaste + Mouthwash | Fluoride Only Toothpaste + Mouthwash
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/61
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days